CLINICAL TRIAL: NCT00237952
Title: Environmental Lead Exposure and Progressive Renal Insufficiency in Patients With Type II Diabetes and Diabetic Nephropathy
Brief Title: Environmental Exposure to Lead and Progressive Renal Insufficiency in Type II Diabetic Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRPG340711; NSC94-2314-B-182A-125
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Diabetic Nephropathies; Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: EDTA chelating agents

SUMMARY:
Background The relationship between long-term heavy lead exposure and chronic interstitial nephropathy is well recognized in the previous literatures. Several epidemiological studies have demonstrated a positive association between blood lead levels and the age related decreases of renal function in the general population and suggested that environmental low-level lead exposure may accelerate the progression of renal function in the healthy persons. In addition, previous our works suggest environmental lead exposure may correlate to progressive renal insufficiency and lead chelation therapy or repeated lead chelation may improve and slow the progressive renal insufficiency in non-diabetic patients with chronic renal diseases. However, Diabetes mellitus is increasing in prevalence worldwide and is currently estimated to affect more than 6.5 percent of the population of the United States. In addition, diabetes is the most common cause of end-stage renal disease in many countries, accounting for about 40 percent of cases. It is still unknown that the relationship between long-term environmental lead exposure and the progressive renal insufficiency in patients with type II diabetes and diabetic nephropathy.

Methods Ninety patints with type II diabetes and diabetic nephropathy (serum creatinine levels between 1.5 mg per deciliter and 3.9 mg per deciliter) who have a normal body lead burden and no history of exposure to lead or other metals will be observed for 24 months. Then, about 50 subjects with high normal body lead burdens (at least 80 μg but less than 600 μg) will be randomly assigned to the study and control groups. For three months, the 25 patients in the study group will receive lead-chelation therapy with calcium disodium EDTA weekly until the body lead burden fallsl below 50 μg, and the 25 control group receive weekly placebo. During the ensuing 12 months, the renal function will be regularly followed up every 3 months and EDTA mobilization tests will be assessed every 6 months. If body lead burden of the study group patients increase more than 60μg, the chelation therapy will be performed again until their body burden are less than 60 μg. The primary end point is an increase in the serum creatinine level to 2 times the base-line value during the observation period. A secondary end point is the change in renal function during the follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 20 through 80 years of age who have type II diabetes mellitus with diabetic nephropathy and followed up at our hospital for more than one year were eligible if they have a serum creatinine concentration between 1.5 mg per deciliter (132.6 μmol per liter) and 3.9 mg per deciliter (344.8 μmol per liter), with a daily proteinuria more than 0.5g/day and no micro-hematuria in urinalysis tests, normal size of both kidneys, retinopathy with laser therapy by ophthalmologists, a history of diabetes more than 5 years and no known history of exposure to lead or other heavy metals (body lead burden, less than 600 μg [2.90 μmol], as measured by EDTA mobilization testing and 72-hour urine collection). Diabetic nephropathy diagnoses are based on the patients' history and the results of laboratory evaluations, renal imaging, and renal histological examination.

Exclusion Criteria:

* type I diabetes; renal insufficiency with a potentially reversible cause, such as malignant hypertension, urinary tract infection, hypercalcemia, or drug-induced nephrotoxic effects; other systemic diseases, such as connective-tissue diseases; use of drugs that may alter the course of renal disease, such as non-steroidal anti-inflammatory agents, steroids, immunosuppressive drugs or Chinese herb drugs.; previous marked exposure to lead (lead poisoning or occupational exposure); drug allergies; and absence of informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-08

PRIMARY OUTCOMES:
The primary end point is an increase in serum creatinine to 1.5 times the base-line value, measured on two occasions one month apart, or the need for hemodialysis during the longitudinal observation period.

SECONDARY OUTCOMES:
A secondary end point is a temporal change in the creatinine clearance or glomerular filtration rate during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Ja-Liang Lin, M.D., Principal Investigator — Chang Gung Memorial Hospital, Lin-Kou Medical Center
Locations (2):
- China (2):
  - Chang Gung Memorial Hospital, Lin-Kou Medical Center, Taipei, Taiwan
  - Chang Gung Memorial Hospital, Taipei, Taiwan